CLINICAL TRIAL: NCT00177619
Title: Prevention of Osteoporosis in Men With Prostate Cancer
Brief Title: Prevention of Osteoporosis in Men With Prostate Cancer on Androgen Deprivation Therapy (POP Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Susan L. Greenspan, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01DK061536 (NIH); 5R01DK061536 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; Bisphosphonates; Hypogonadism
MeSH Terms: conditions — Prostatic Neoplasms; Hypogonadism | interventions — Alendronate

INTERVENTIONS:
Drug: Alendronate

SUMMARY:
The overall goal of this proposal is to determine the effectiveness and safety of once weekly alendronate (Fosamax) in the prevention and treatment of osteoporosis in men with prostate cancer on androgen deprivation therapy and to evaluate maintenance of bone mass following termination of therapy after one year.

DETAILED DESCRIPTION:
While osteoporosis in women is recognized as a major public health problem, osteoporosis in men also has a profound clinical impact. Men over the age of 75 who sustain hip fractures have a higher mortality than women of the same age (30% versus 9%). Hip fractures in men account for one-third of all hip fractures. In 1995, male osteoporosis accounted for $2.7 billion in health care costs -- nearly one-third of the overall cost of osteoporosis. Alendronate has been shown to improve bone mass and decrease vertebral fractures in men with osteoporosis.

Prostate cancer is the most common visceral malignancy and the second leading cause of death in American men. Almost all men who progress to late stage disease are treated with androgen deprivation therapy for life, resulting in a 5-fold increased risk of hip fractures and a 13-fold increased risk of all osteoporosis fractures. Several studies suggest the merit of inducing androgen deprivation much earlier in the course of therapy for prostate cancer. It is therefore quite likely that androgen deprivation strategies will be employed with increasing frequency in patients with less advanced disease, resulting in longer life expectancy but greater bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18 and older with stage Do prostate cancer (as defined by asymptomatic disease, rising PSA, and negative bone scans) following attempted curative surgery and/or radiation
* Androgen deprivation therapy (gonadotropin releasing hormone agonists, lutenizing hormone releasing hormone agonists, testosterone antagonists, orchiectomy) for at least 6 months for treatment of prostate cancer

Exclusion Criteria:

* History of any illness known to affect bone and mineral metabolism (renal failure, hepatic failure, Paget's disease, osteogenesis imperfecta, osteomalacia)
* Non-prostate cancer diagnosed within last 5 years (treated superficial basal and squamous cell carcinoma excepted)
* Hyperparathyroidism
* Malabsorption
* Treatment with medications known to affect bone metabolism (chronic high-dose corticosteroid therapy for at least 6 months, thyroid hormone with TSH <0.1 micrograms, antiseizure medications)
* Active peptic ulcer
* Inability to sit upright or stand for at least 30 minutes
* Kidney stones in the past 5 years
* 24-hour urine calcium value >400 mg/24 hours
* Esophageal stricture or achalasia
* Hyperthyroidism
* Evidence of chronic liver disease (including alcoholism)
* Treatment within past year for osteoporosis (calcitonin, fluoride, bisphosphonates)
* History of atraumatic fractures, previous fracture due to a fall from standing height or lesser trauma, or clinical osteoporosis
* Metastatic prostate cancer
* Inability to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Our primary outcome variable will be change in spine bone mineral density over one year and change during the second year (or both years).

SECONDARY OUTCOMES:
Secondary endpoints will be bone mineral density at the hip and lateral spine.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States